CLINICAL TRIAL: NCT04711798
Title: Study of Perioperative Evolution of Right Heart Dysfunction and Preload Responsiveness in Open Heart Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN172020/CHUSTE
Record Dates: First submitted 2021-01-05; First posted 2021-01-15 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Surgery
Keywords: Lung recruitment maneuver; Fluid responsiveness; cardiac surgery; right cardiac dysfunction; passive leg raising; Transcardiopulmonary Thermodilution; Calibrated Arterial Waveform Analysis; echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving cardiac surgery: Patients receiving cardiac surgery will be included. All patients received a passive leg raising maneuver (PLR) for preload status evaluation using the PICCO system, a lung recruitment maneuver (LRM) and an echographic evaluation of the right cardiac function.
  Interventions: Other: passive leg raising maneuver (PLR); Other: lung recruitment maneuver (LRM); Other: echographic evaluation of the right cardiac function

INTERVENTIONS:
Other: passive leg raising maneuver (PLR) — Passive leg raising maneuver (PLR) for preload status evaluation using the PICCO system will be realized in Phase 1 (pre operatively), Phase 2 (after the sternotomy closure in the operating room), Phase 3 (H+2 of the arrival in cardiac intensive care unit).
Other: lung recruitment maneuver (LRM) — lung recruitment maneuver (LRM) will be realized in Phase 1 (pre operatively), Phase 2 (after the sternotomy closure in the operating room), Phase 3 (H+2 of the arrival in cardiac intensive care unit).
Other: echographic evaluation of the right cardiac function — echographic evaluation of the right cardiac function will be realized in Phase 1 (pre operatively), Phase 2 (after the sternotomy closure in the operating room), Phase 3 (H+2 of the arrival in cardiac intensive care unit).

SUMMARY:
The aim of the study was to assess the ability a Lung Recruitment Maneuver (LRM) with a stepwise increase of PEEP to predict fluid responsiveness and right cardiac dysfunction in mechanically ventilated patients in open heart cardiac surgery. During different phases, all patients received a Passive Leg Raising (PLR) maneuver for preload status evaluation using the PICCO system, a Lung Recruitment Maneuver (LRM) and an echographic evaluation of the right cardiac function. 20 patients were analyzed. Incomplete Lung Recruitment Maneuver (LRM) can predict fluid responsiveness at phase 1, pre-operatively, with a sensitivity of 0.57 and specificity of 0.62. Performance of an incomplete Magnetic Resonance Angiography (MRA) to predict right cardiac dysfunction based on TAPSE post-operatively provides a sensitivity and specificity of respectively 0.33 and 0.17 Tolerance to a stepwise lung recruitment maneuver can not be used to evaluate reliably the preload responsiveness and guide fluid therapy except pre-operatively. The use of a lung recruitment maneuver can be a promising method for right cardiac dysfunction screening but further studies need to be done with different echographic tools for right cardiac dysfunction evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving an elective or urgent cardiac surgery with or without extracorporeal circulation under general anesthesia, under protective mechanical ventilation, monitored by invasive arterial blood pressure and pulse contour analysis (PICCO system) for cardiac output measurement and central venous pressure

Exclusion Criteria:

* Left ventricular ejection fraction ≤ 30%
* heart arrhythmia, pulmonary hypertension (SPAP > 35 mmHg)
* right heart failure (TAPSE < 16 mm, S' at lateral tricuspid valve < 10 cm/sec)
* lower limbs obstructive arteriopathy (stage IIb, III and IV)
* severe and very severe chronic obstructive pulmonary disease (COPD)
* pneumothorax and extreme weights (BMI < 35 kg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receive cardiac surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness measured with PiCCO system during Lung recruitment maneuver. | Months: 4
  Measured by PICCO results (phase: 1, 2, 3).

SECONDARY OUTCOMES:
Analysis Right cardiac function - Transthoracic echocardiography | Months: 4
  measured with Transthoracic echocardiography (phase 1, 3).
Analysis Right cardiac function - transoesophageal echocardiography | Months: 4
  measured with transoesophageal echocardiography (phase 1, 2).

CONTACTS AND LOCATIONS:
Overall Officials: Camille BELLOT, resident, Study Chair — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No